CLINICAL TRIAL: NCT00875745
Title: Phase I, Open-label, Dose-escalation Study of the Combination of Sorafenib and Vorinostat in Poor-risk Acute Myelogenous Leukemia (AML) and High Risk Myelodysplastic Syndrome (MDS)
Brief Title: Combination of Sorafenib and Vorinostat in Poor-risk Acute Myelogenous Leukemia (AML) and High Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0902-08; IUCRO-0234
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute; Myelodysplastic Syndromes | interventions — Sorafenib; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib-Vorinostat (Experimental): This is a single-arm, non-randomized feasibility and safety Phase I trial of a combination of Sorafenib and Vorinostat, both administered orally.
  Interventions: Drug: Sorafenib-Vorinostat

INTERVENTIONS:
Drug: Sorafenib-Vorinostat — Patients will be entered in successive cohorts. The first cohort will receive Sorafenib at 400 mg bid (800 mg daily) and Vorinostat at 100 mg bid (200 mg daily).
  Other Names: Nexavar (Sorafenib); Zolinza (Vorinostat)

SUMMARY:
The purpose of this study is to test the safety of sorafenib and vorinostat when given together to see what effects (good and bad) it has on the patient and their acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS). This study is also being done to find the highest dose of sorafenib and vorinostat that can be given together without causing severe side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of AML (> 20% myeloid blasts in the peripheral blood or bone marrow) or MDS with > 10% myeloid blasts in the bone marrow. Patients with Acute Promyelocytic Leukemia (APL) must be refractory to all-trans retinoic acid (ATRA) and arsenic trioxide.
* The patients must have one of the following criteria:

  * Age of 18 to 69 years; relapsed or refractory disease following at least one prior therapeutic regimen; not a candidate for cytotoxic or other conventional therapies due to disease refractoriness, poor performance status, or co-morbidities
  * Age of 70 years or older; received no previous therapies (other than hematopoietic growth factors or hydroxyurea); not a candidate for cytotoxic or other conventional therapies due to poor performance status, co-morbidities, or personal preference
  * Age of 70 years or older with relapsed or refractory disease
* The patient must have discontinued all previous therapies for acute leukemia for at least 14 days and recovered from the acute effects of the therapy.
* Patients must have an ECOG (Zubrod) performance status of 0-2
* Patients must be able to take and tolerate oral medications
* Patients must have adequate organ function as specified in the protocol.
* Patients not on anti-coagulation must have an INR < 1.5 and a PTT within normal limits.

Exclusion Criteria:

* Pregnant women or nursing mothers are not eligible for this trial.
* Patients may receive no other concurrent biologic therapy, cytotoxic chemotherapy or radiation therapy during this trial.
* Patients with one or more serious preexisting medical conditions that, in the opinion of the investigator, would preclude participation in this study. See protocol for listing.
* Patients with known central nervous system (CNS) leukemia by spinal fluid cytology, flow cytometry or imaging
* Patients with previous autologous or allogeneic stem cell transplantation who have current side effects and/or complications that in the opinion of the investigator can interfere with the interpretation of the toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of a combination of Sorafenib and Vorinostat administered to patients with poor-risk AML, or MDS with >10% blasts. | Baseline through cycle 3

SECONDARY OUTCOMES:
Evaluate response and the duration of response to this combination targeted therapy | Baseline through Cycle 3
Evaluate the toxicity of the combination of Sorafenib and Vorinostat in patients receiving this therapy | Baseline through Cycle 3

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Sayar, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States